CLINICAL TRIAL: NCT06602375
Title: The Effect of Manual Physical Therapy and Exercise in Addition to Routine Dental Care in Individuals With Temporomandibular Disorders: a Randomized Controlled Trial
Brief Title: The Effect of Manual Physical Therapy and Exercise in Addition to Routine Dental Care in Individuals With Temporomandibular Disorders
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Brooke Army Medical Center (U.S. Federal Agency)
Responsible Party: Principal Investigator, Mason A Frank, Physical Therapist, Brooke Army Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: C.2024.090d; 974205 (Other: San Antonio Institutional Review Board, Brooke Army Medical Center, Defense Health Agency)
Record Dates: First submitted 2024-09-16; First posted 2024-09-19 (Actual); Last update posted 2025-02-05 (Actual); Status verified 2024-09

CONDITIONS: Temporomandibular Disorders (TMD)
Keywords: Temporomandibular Disorders; Physical Therapy; Manual Therapy; Exercise
MeSH Terms: conditions — Temporomandibular Joint Disorders; Motor Activity | interventions — Standard of Care; Physical Therapy Modalities

STUDY DESIGN:
Intervention Model Description: This study will be a pragmatic, parallel randomized controlled trial. Participants will be randomly assigned to either the experimental (standard care plus physical therapy) or control (standard care) group.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Standard care plus physical therapy (Experimental): Participants randomized to this group will receive standard care from their treating dental provider. In addition, they will receive routine physical therapy interventions over a 6-week (+/- 2 week) period. Study participants will receive treatments based on their clinical examination. Subjects will attend up to 12 sessions over 6-weeks (+/- 2 weeks). The initial physical therapy visit will be 60-minutes long with all subsequent appointments being 30-minutes, to include any booster sessions. The interventions will be pragmatic in nature, with provided treatment being specific to the subject's specific complaints, goals, and examination identified impairments.
  Interventions: Other: Standard care; Other: Physical Therapy (PT)
- Standard Care (Active Comparator): Those randomized to the standard care (control) group will follow the plan of care determined by their treating dental provider. This group will receive standard (routine) care from the dental provider for the treatment of TMD. These decisions will be based on the clinical judgment of the dental provider, as is customary with routine care for TMD.
  Interventions: Other: Standard care

INTERVENTIONS:
Other: Standard care — The standard care (control) group will follow the plan of care determined by their treating dental provider. These decisions will be based on the clinical judgment of the dental provider and subject desires. Intervention may include, but is not limited to typical patient education, pharmacotherapy, oral splinting or occlusal device, cryo/thermotherapy recommendations, and exercise handouts.
Other: Physical Therapy (PT) — Participants randomized to this group will receive individualized, tailored courses of physical therapy care. Interventions may be directed at the temporomandibular, cervical, and/or scapulothoracic regions based on subject clinical presentation and impairments. Manual therapy joint and soft tissue mobilizations may be used to address pain, mobility, and motor control. Motor control exercises may be used to promote relaxation, improve range of motion, and appropriate postures. Strengthening exercise, primarily directed to the cervical and scapulothoracic regions, may be implemented as appropriate. Stretching exercise may be used to address pain and mobility deficits. The interventions are intentionally pragmatic; study participants will receive treatment as they are comfortable and as recommended by the treating therapist.
  Arms: Standard care plus physical therapy

SUMMARY:
The goal of this randomized clinical trial among US military active-duty service-members with temporomandibular disorders (TMD) is to determine whether standard care plus 6-weeks of tailored, individualized physical therapy (PT) treatment provides greater benefit than standard care alone in patient-reported outcomes, and maximal mouth opening.

The aims of the study are to compare outcomes in individuals with TMD that receive standard care treatment versus standard care plus PT interventions at 0-, 6-, and 12-weeks. The investigators anticipate that subjects in the standard care plus PT group will exhibit improved patient-reported outcomes, and maximal mouth opening compared to those who received standard care alone.

Additionally, the investigators will compare the amount and type of healthcare utilization between the two groups (Standard Care and Standard Care + PT) in the 12-month period following enrollment in the study.

All participants will be managed by their primary dental provider and receive care as deemed appropriate by their provider. All participants will complete patient-reported outcome measures and have their jaw motion measured. Those randomized to the standard care plus PT group will also receive a tailored PT evaluation followed by an individualized plan of care two times per week for up to six weeks.

DETAILED DESCRIPTION:
The following procedures will be conducted once the subject has signed and received their informed consent and Health Insurance Portability and Accountability Act (HIPAA) documents.

Inclusion/exclusion will be reviewed (including the TMD Pain Screener). Subjects will then be provided with research questionnaires and patient-reported outcome measures for completion. All outcomes will be obtained through direct interaction with subjects.

Subjects will then undergo measurements for pain-free mouth opening and maximal mouth opening (MMO) ranges of motion. All subjects will undergo the same measurement protocol.

Following the above measures, subjects will then be randomized into one of two parallel treatment arms, standard care (control group), or standard care + PT interventions (experimental group). The groups are further described below. The method of group assignment will be sequentially numbered opaque sealed envelopes (SNOSE). To minimize the risk of predicting the treatment assignment of the next eligible subject, randomization will be performed in permuted blocks of 2 or 4 with random variation of the blocking number. Due to the nature of the study, it is not possible to blind the subjects or the clinician providing the intervention to the treatment received. Assessors will be blinded to group allocation, and clinicians will be blinded to outcomes.

After randomization, enrolled subjects who have already received care from a dental provider will continue with their dental provider for routine TMD care. Any enrolled subjects not being seen by a dental provider for their TMD concerns will be referred to the prosthodontist associated with this study.

These enrollment procedures may last up to one hour.

Those randomized to the standard care (control) group will follow the plan of care determined by their treating dental provider. This group will receive standard (routine) care from the dental provider for the treatment of TMD. These decisions will be based on the clinical judgment of the dental provider, as is customary with routine care for TMD.

Participants randomized to the standard care + PT interventions (experimental) group will receive standard care from their treating dental provider. In addition, they will receive routine physical therapy interventions over a 6-week (+/- 2 week) period. Study participants will receive treatment based on their clinical examination, as is typical for routine physical therapy clinical practice. Subjects will attend up to 12 sessions over 6-weeks (+/- 2 weeks), as is typical for physical therapy management of TMD conditions. The initial physical therapy visit will be 60-minutes long with all subsequent appointments being 30-minutes, to include any booster sessions.

The interventions will be pragmatic in nature, with provided treatment being specific to the subject's specific complaints, goals, and examination identified impairments, as is customary for physical therapist management of TMD conditions. Physical therapists will progress the program at the rate perceived to be most efficacious for the participant's needs. All PT interventions utilized in this study are considered routine care for individuals with TMD.

This study is intentionally pragmatic in that study participants will receive treatment as they are comfortable and as recommended by the treating providers. For example, it is not expected that every patient receives cervical spine mobilizations during physical therapy, however in some of the participants this may be needed to aid in beneficial treatment. Similarly, dental providers are not required to provide splinting or medications to all participants. Provided treatment will be based on providers clinical reasoning as it customary.

Both groups will have follow-up outcomes collected at 6-weeks (+/- 3 days) following study enrollment. All outcomes will be obtained through direct interaction with subjects.

Between the 6- and 12-week data collection appointments all subjects may continue with standard care interventions and processes as indicated and recommended by the overseeing dental provider. Subjects assigned to the experimental group will have the option of booster treatment sessions with one of the research team members. Booster sessions refer to the subject choosing to attend more appointments after their course of care has been completed, should their symptoms return. In this case, booster sessions would be available between the 6 and 12-week follow-up time points. Booster sessions will be limited to two sessions as is typical with physical therapy practice. Booster sessions will last 30-minutes and are routinely offered for patients at the participating Physical Therapy Clinic as part of typical clinical practice for physical therapy management of musculoskeletal conditions.

Both groups will have follow-up outcomes collected at 12-weeks (+/- 3 days) following study enrollment.

Subjects enrolled in the standard care only group, who are not satisfied with their clinical progress, will be offered physical therapy services at this time. This care will be unrelated to study aim 1 of this research and no additional data collection will occur.

Healthcare utilization data will be collected from the Military Health System Data Repository (MDR) database and will be confirmed via electronic health record system review. Healthcare utilization data will be used to determine any subsequent medical utilization related to TMD. To collect this information a Data Sharing Agreement (DSA) will be completed between the research team and the Defense Health Agency (DHA). A signed, completed IRB protocol is required prior to submitting the DSA. However, this should not impact the timing of this study as the data pull will be completed after the last enrolled subject's final follow-up at 12-weeks post-enrollment. This will provide enough time to complete the data sharing agreement (DSA) with both agencies before performing this analysis. Details for determining the health care utilization are outlined below:

The goal of the MDR database will be to determine which of these subjects sought health care related to TMD in the 12-month period after treatment in this study. This data will allow us to determine the extent of healthcare utilization incidence in both groups.

Recording of Extracted Data with Identifiers: The data will be provided in a coded manner from the data analysts. These analysts are Defense Health Agency (DHA) employees with full authorized access to these Department of Defense (DoD) databases. They must have a signed Data Sharing Agreement from the Privacy Board of the DHA to pull the requested data. They have full authorization to access and pull this data, as they do this regularly for business operations and operational decision making by leaders at the DHA. As they have done before with members of our team on prior projects, they extract all the required data based upon the name, age, and DoD identification number that the Research Team provides to the analyst to identify the correct subjects that were in the study. Investigators will see the provided PII (via secure safe AMRDC or encrypted government email) as they need this for the extraction. However, they will replace everything with a pseudo identification number that aligns with the study subject ID before returning the coded (de-identified) data back to the research team for analysis. Before any personal identifying information (PII) is released, each research subject will authorize the release through a signed HIPAA Authorization Document. The analyst will also assign a pseudo identification number matched with the list of our subject PHI that the investigators provided to them. Therefore, the final working set they provide us for analysis will not have any identifying PHI/PII associated with it. If additional follow-up is needed to clarify a health care utilization event in MHS GENESIS, the research team can check the master subject record (stored by the PI on an encrypted computer) to link the pseudo identification number to DOD ID. Therefore, prior to analysis occurring, only files with coded identifiers will be used. Confidentiality of protected health information will always be maintained by the PI. The final working database to be used in the data analysis will not include PHI information.

Location of Extracted and Recorded Data: The health care utilization data will be extracted from the MDR database. Even though the data is now coded, the extracted data will still be maintained in an encrypted, password protected file kept at the participating physical therapy clinic, Brooke Army Medical Center by the PI. All data collection forms, and the master participant list will be secured in an office at the participating physical therapy clinic. All data maintained on a computer will be password protected and only accessible by the study investigators.

Nature of Identifying Data: Timeframes will be requested in reference to the baseline enrollment date rather than the actual date of the visit. For example, the date of appointment will be required initially to determine when the healthcare visit associated with the TMD occurred. However, this data will be coded differently in the working spreadsheet. Data will be returned with the days from the index date (enrollment) listed rather than a date. For example, a subject was enrolled on 1 Jun 2024 and then had a medical visit of interest on 15 July 2024. The encounter will be +45 as an indicator of the visit occurring 45 days after enrollment. Analysis of the data will only occur in the coded spreadsheet that will not have dates.

Status of the extracted data after completion of the research study: At the study completion, the Master Key file linking the participant's PII to the study will be deleted. The PI will then provide an electronic copy of the most current version of the protocol, IRB approval letter, final report, signed HIPAA Authorizations and the most current version of the ICD for indefinite archiving. The PI will submit a copy of all ICD signature pages as well. An electronic copy of all signed HIPAAs and ICDs will be provided to the Protocol Office during each Progress Report submittal. After at least six years, the data will be destroyed in accordance with research department protocol. Full compliance with Health Insurance Portability and Accountability Act (HIPAA) standards will be upheld throughout the investigation to protect confidentiality.

ELIGIBILITY:
Inclusion Criteria:

* Active-Duty Service Members
* Complaint of TMD symptoms
* Must be able to be followed for twelve weeks after consent
* TMD Screener score ≥ 3 45

Exclusion Criteria:

* Actively in a Trainee status
* Utilized oral device in past 6 months
* Facial injection therapy in the prior 6 months
* Facial surgery in the preceding 6 months
* Serious spinal pathology (acute fracture, active cancer, instability)
* Diagnosed neurological or rheumatological disease
* Currently under litigation related to temporomandibular or cervical spine pain(s)
* Currently undergoing Medical Evaluation Board (MEB)
* Retiring or separating from the military within a year

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-09-16 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Jaw Functional Limitation Scale - 8 item (JFLS-8) | From enrollment to 12 weeks post enrollment (primary), will also be assed at 6-weeks
  This study's primary outcome variable is the Jaw Functional Limitation Scale - 8 Item version. This 8-item questionnaire is scored from 0 to 80 points, with higher scores indicating greater levels of functional limitation. The JFLS-8 is a reliable and valid tool to measure patient functional limitations related to the jaw. This questionnaire is supported by the dental and physical therapy communities to measure functional limitations of the jaw. Each item is scored from 0-10. The scores are summed and divided by the number of items answered. No more than two items can be missing for scoring to take place.

SECONDARY OUTCOMES:
Numeric Pain Rating Scale (NPRS) | At enrollment, 6-weeks, and 12-weeks
  The Numeric Pain Rating Scale is an 11-point scale from 0-10 that measures pain intensity in adults, with higher scores indicating greater levels of pain. Subjects will select a value that is most in line with their current perceived pain intensity. The NPRS is a reliable and valid tool. The minimal clinically important difference has been widely established as two points.
Neck Disability Index (NDI) | Collected at baseline, 6- and 12-weeks.
  The Neck Disability Index (NDI) contains 10-items scored from 0-5 on a Likert scale which assesses the construct of neck related disability. Scores range from 0 to 50 and are reported as percentages, with higher scores associated with greater levels of disability. The NDI is a valid, reliable, and responsive tool with a minimal clinically importance difference reported as 7.5 points, or 15%.
Central Sensitization Inventory (CSI) | Collected at baseline, 6- and 12-weeks.
  The Central Sensitization Inventory (CSI) is a reliable and valid 25-item questionnaire with each item assessed on a scale ranging from "never" (0 points) to "always" (4 points) with a resultant score between 0 and 100. Scores higher than 40 points are suggestive of a central sensitization component to patient symptoms. This score will be dichotomized with scores of 40 or higher indicating central sensitization, and scores of 39 or less indicating no presence of central sensitization.
Global Rating of Change (GRoC) | Collected at 6- and 12-weeks
  The Global Rating of Change (GRoC) scale is a valid measure of a patient's overall perceived change in quality of life through an 11-point Likert scale. The scale ranges from "-5" to "+5" associated with "very much worse" to "completely recovered," respectively. The minimal clinically important difference is a change greater than or equal to two points. This score will be dichotomized with scores 3+ or greater indicating improvement, and scores 2 or less indicating no improvement.
Pain-Free Mouth Opening (PFMO) | Collected at baseline, 6- and 12-weeks.
  Pain-free maximal mouth opening (PFMO) is an important clinical measure that has implications for a subject's ability to talk and eat. This is measured in millimeters between the upper and lower central incisors via a standard single-use, disposable jaw range of motion assessment tool. Three trials at each time point will be performed, and the average utilized for statistical analysis. A meaningful change in this range of motion has not been established, however 40mm is widely considered a normal range of motion. Measures will be reported to the nearest millimeter.
Maximal Mouth Opening (MMO) | Collected at baseline, 6- and 12-weeks
  Maximal mouth opening (MMO) is an important clinical measure that has implications for a subject's ability to talk and eat. This is measured in millimeters between the upper and lower central incisors via a standard single-use, disposable jaw range of motion assessment tool. Three trials at each time point will be performed, and the average utilized for statistical analysis. A meaningful change in this range of motion has not been established, however 40mm is widely considered a normal range of motion. Measures will be reported to the nearest millimeter.
Healthcare Utilization | Collected at 12-months after enrollment for each subject
  Healthcare utilization data will be collected from the MHS Data Repository (MDR) database and will be confirmed via MHS GENESIS. Healthcare utilization data will be used to determine any subsequent medical utilization related to TMD. This data will include type of healthcare utilized, location of healthcare, number of clinic visits, types of specialty clinics visited, associated imaging, associated medication, associated procedures/surgeries, and current procedural terminology (CPT) codes.
Patient-Report Outcome Measure Information System (PROMIS-57) | Collected at baseline, 6- and 12-weeks.
  The Patient-Report Outcome Measure Information System-57 (PROMIS-57) is a patient-reported outcome measure developed by the National Institute of Health. It is a universal measure that assesses physical, mental, and social health across diverse conditions, to include orthopedic conditions. The PROMIS-57 questions cover seven health domains: physical function, anxiety, depression, fatigue, sleep disturbance, social participation, and pain. These domains have been less extensively studied in the orofacial pain population, but changes of 2-6 T-score points are reasonable estimates for MCID across domains. In the physical function and social participation domains, higher scores are representative of greater function and participation, respectively. In the domains of pain interference, fatigue, sleep disturbance, anxiety, depression, and pain intensity, lower scores are associated with lower impact of the associated construct.

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin R Hando, PhD, DPT, Study Chair — Army-Baylor Doctoral Fellowship in Orthopedic Manual Physical Therapy, Brooke Army Medical Center
Locations (1):
- Brooke Army Medical Center, Fort Sam Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No
Requests for deidentified data will be considered on a case-by-case basis.

REFERENCES:
- [Background] Valesan LF, Da-Cas CD, Reus JC, Denardin ACS, Garanhani RR, Bonotto D, Januzzi E, de Souza BDM. Prevalence of temporomandibular joint disorders: a systematic review and meta-analysis. Clin Oral Investig. 2021 Feb;25(2):441-453. doi: 10.1007/s00784-020-03710-w. Epub 2021 Jan 6. PMID 33409693
- [Background] Fernandez-de-Las-Penas C, Von Piekartz H. Clinical Reasoning for the Examination and Physical Therapy Treatment of Temporomandibular Disorders (TMD): A Narrative Literature Review. J Clin Med. 2020 Nov 17;9(11):3686. doi: 10.3390/jcm9113686. PMID 33212937
- [Background] von Piekartz H, Schwiddessen J, Reineke L, Armijo-Olivio S, Bevilaqua-Grossi D, Biasotto Gonzalez DA, Carvalho G, Chaput E, Cox E, Fernandez-de-Las-Penas C, Gadotti IC, Gil Martinez A, Gross A, Hall T, Hoffmann M, Julsvoll EH, Karegeannes M, La Touche R, Mannheimer J, Pitance L, Rocabado M, Strickland M, Stelzenmuller W, Speksnijder C, van der Meer HA, Luedke K, Ballenberger N. International consensus on the most useful assessments used by physical therapists to evaluate patients with temporomandibular disorders: A Delphi study. J Oral Rehabil. 2020 Jun;47(6):685-702. doi: 10.1111/joor.12959. Epub 2020 May 4. PMID 32150764
- [Background] Bhargava D, Chavez Farias C, Ardizone Garcia I, Mercuri LG, Bergman S, Anthony Pogrel M, Sidebottom AJ, Srouji S, Senturk MF, Elavenil P, Moturi K, Anantanarayanan P, Bhargava PG, Singh VD. Recommendations on the Use of Oral Orthotic Occlusal Appliance Therapy for Temporomandibular Joint Disorders: Current Evidence and Clinical Practice. J Maxillofac Oral Surg. 2023 Sep;22(3):579-589. doi: 10.1007/s12663-023-01939-y. Epub 2023 Jun 27. PMID 37534353
- [Background] Orzeszek S, Waliszewska-Prosol M, Ettlin D, Seweryn P, Straburzynski M, Martelletti P, Jenca A Jr, Wieckiewicz M. Efficiency of occlusal splint therapy on orofacial muscle pain reduction: a systematic review. BMC Oral Health. 2023 Mar 28;23(1):180. doi: 10.1186/s12903-023-02897-0. PMID 36978070
- [Background] Cella D, Choi SW, Condon DM, Schalet B, Hays RD, Rothrock NE, Yount S, Cook KF, Gershon RC, Amtmann D, DeWalt DA, Pilkonis PA, Stone AA, Weinfurt K, Reeve BB. PROMIS(R) Adult Health Profiles: Efficient Short-Form Measures of Seven Health Domains. Value Health. 2019 May;22(5):537-544. doi: 10.1016/j.jval.2019.02.004. PMID 31104731
- [Background] DeSouza CM, Legedza AT, Sankoh AJ. An overview of practical approaches for handling missing data in clinical trials. J Biopharm Stat. 2009 Nov;19(6):1055-73. doi: 10.1080/10543400903242795. PMID 20183464
- [Background] Hoffmann RG, Kotchen JM, Kotchen TA, Cowley T, Dasgupta M, Cowley AW Jr. Temporomandibular disorders and associated clinical comorbidities. Clin J Pain. 2011 Mar-Apr;27(3):268-74. doi: 10.1097/AJP.0b013e31820215f5. PMID 21178593
- [Background] Idanez-Robles AM, Obrero-Gaitan E, Lomas-Vega R, Osuna-Perez MC, Cortes-Perez I, Zagalaz-Anula N. Exercise therapy improves pain and mouth opening in temporomandibular disorders: A systematic review with meta-analysis. Clin Rehabil. 2023 Apr;37(4):443-461. doi: 10.1177/02692155221133523. Epub 2022 Oct 20. PMID 36263523
- [Background] Asquini G, Pitance L, Michelotti A, Falla D. Effectiveness of manual therapy applied to craniomandibular structures in temporomandibular disorders: A systematic review. J Oral Rehabil. 2022 Apr;49(4):442-455. doi: 10.1111/joor.13299. Epub 2022 Jan 17. PMID 34931336
- [Background] Minervini G, Franco R, Marrapodi MM, Fiorillo L, Cervino G, Cicciu M. Post-traumatic stress, prevalence of temporomandibular disorders in war veterans: Systematic review with meta-analysis. J Oral Rehabil. 2023 Oct;50(10):1101-1109. doi: 10.1111/joor.13535. Epub 2023 Jun 23. PMID 37300526